# **Informed Consent Form**

Official Title: Comparison of Total Intravenous Anesthesia Methods in Patients Undergoing

Neuromonitoring

**NCT Number:** Pending (Not yet assigned)

**Document Date:** May 10, 2023

#### INFORMED CONSENT FORM

**DOCUMENT NO:** EY.FR.050 **PUBLICATION DATE:** 30.01.2019

**REVISION DATE/REVISION NO: 00/00** 

### Comparison of Total Intravenous Anesthesia Methods in Spinal Surgery

This form aims to provide information about the study you are invited to participate in and to obtain your consent for participation.

The study titled "Comparison of Total Intravenous Anesthesia Methods in Spinal Surgery" will be conducted with voluntary participants by Dr Ayşegül DANACI. The study aims to demonstrate that intraoperative limited opioid consumption achieved with different total intravenous anesthesia methods can lead to reduced postoperative opioid analgesic requirements, lower pain scores, and decreased hyperalgesia incidence. The expected duration of participation in this study is 24 hours.

From May 15, 2023, a total of 72 volunteers will be included in the study. Patient history, the doses of drugs used during the maintenance of anesthesia, BIS range, pain assessment, and postoperative analgesic needs will be recorded for the patients participating in the study. The study will be conducted at the **Dr. Abdurrahman Yurtaslan Oncology Training and Research Hospital.** 

Your participation in the study is voluntary. The information obtained during the study will be kept confidential, will not be disclosed to the public, and even if the results of the study are published, your identity will remain anonymous and will only be used for research purposes. However, the study investigator, ethics committee, institution, and other relevant health authorities may have direct access to your medical records. At the end of the study, you have the right to request infor

mation about your results. By signing the written informed consent form, you or your legal representative will grant permission for such access.

If new information is obtained during the study that may affect your willingness to continue participating, you or your legal representative will be promptly informed.

For any questions or concerns regarding the study, you may contact **Dr. Ayşegül DANACI** at +90 5541362515 at any time, 24/7. You have the right not to participate in this study. After agreeing to participate, you may withdraw from the study at any stage without any penalty or repercussions. Additionally, the investigator may exclude you from the study if deemed necessary. In cases of non-participation, withdrawal, or exclusion, there will be no penalties

or loss of any benefits to which you are entitled. This study is conducted solely for research purposes, and no experimental drug testing will be carried out. The treatment plan devised by your treating physician will not be altered during this study.

If you participate in this study, no payment will be made to you, and no fees will be charged. This study is not sponsored by any institution or organization. Approving this form means you consent to participate in the study.

# **Participation Approval:**

I have read and listened to the information provided above, which must be given to the volunteer before the study begins. I have asked all the questions that came to my mind to the investigator, and I fully understand all the written and verbal explanations made to me. I was given sufficient time to decide whether I wanted to participate in the study. Under these conditions, I authorize the research investigator to review, transfer, and process my medical information, and I voluntarily accept the invitation to participate in the study without any coercion or pressure.

A signed copy of this form will be given to me.

| Volunteer: |
|-------------------|
| Name and Surname: |
| Date: |
| Signature: |

### Legal Representative/Guardian/Relative of the Volunteer:

Name and Surname:
Date:
Signature:

# **Investigator:**

Name and Surname: Date:

Signature:

## Witness:

Name and Surname:

Date:

Signature: